CLINICAL TRIAL: NCT03699709
Title: Cooking for Health in a Large American Indian Community in the North-Central United States
Brief Title: Cooking for Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Medstar Health Research Institute (Other); Missouri Breaks Industries Research, Inc. (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Amanda Fretts, Assistant Professor, School of Public Health: Epidemiology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00004114; R01MD011596 (NIH)
Record Dates: First submitted 2018-10-02; First posted 2018-10-09 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diet; cooking skills
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Budgets

STUDY DESIGN:
Intervention Model Description: Randomization to one of two arms: intervention or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental)
  Interventions: Behavioral: Budgeting, purchasing and cooking educational intervention
- Control Arm (No Intervention)

INTERVENTIONS:
Behavioral: Budgeting, purchasing and cooking educational intervention — Receive culturally-tailored healthy food budgeting, purchasing, and cooking skills curriculum
  Arms: Intervention Arm

SUMMARY:
Type 2 diabetes is a leading cause of morbidity and mortality among American Indians (AIs) in the United States. Although healthy diet is a key component of diabetes management programs, many AIs face barriers to adopting a healthy diet including: difficulty budgeting for food on low-incomes, low literacy and numeracy when purchasing food, and limited cooking skills. The proposed project will evaluate a culturally-targeted healthy foods budgeting, purchasing, and cooking skills intervention aimed at improving the cardio-metabolic health of AIs with type 2 diabetes who live in rural areas.

DETAILED DESCRIPTION:
The research activities proposed in this application address a pressing need in American Indian (AI) communities - the evaluation of a culturally-tailored healthy food budgeting, purchasing, and cooking intervention to see whether it can improve diet and health among AIs with type 2 diabetes.

This randomized clinical trial will compare the efficacy of a culturally-tailored healthy food budgeting, purchasing, and cooking program on: (1) diet quality (i.e., intake of sugar-sweetened beverages, processed foods) and (2) healthy food budgeting and cooking skills, among AIs with type 2 diabetes who reside in a large AI community in the north-central United States. Additionally, the investigators will conduct a mixed methods process evaluation to assess intervention reach, fidelity, and participant satisfaction. Curriculum will be tailored to an AI population with diabetes, and directly address major barriers to healthy eating that were identified by community members and tribal leaders in recent focus groups including: (1) difficulty budgeting for food on low-incomes; (2) low literacy and numeracy when purchasing food (e.g., inability to use in-store scales to convert foods priced "per pound" to dollar values); (3) limited cooking skills. The investigators expect that implementation of a culturally-tailored diet intervention will be effective in promoting positive diet change, and increase healthy food budgeting and cooking skills.

Poorly controlled diabetes affects the health/longevity of those afflicted, and has profound effects on healthcare costs. Greater efforts are needed to encourage healthy eating in underserved communities with a high burden of diabetes. Improving healthy food budgeting, purchasing, and cooking skills among AIs with diabetes should improve diet and diabetes management. If successful, this program can be extended to other AI communities.

ELIGIBILITY:
Inclusion Criteria:

* American Indian
* 18+ years
* self-reported type 2 diabetes
* reside on reservation where study is being conducted
* self-identify as person who holds most of the responsibility for household budgeting, shopping, and cooking

Exclusion Criteria:

* pregnant
* history of bariatric surgery
* chronic kidney disease
* on dialysis
* cognitively impaired
* individuals without a reliable place to cook or store food (e.g., homeless)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2023-11-26 (Actual); Study Completion 2023-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda M Fretts, PhD, Principal Investigator — University of Washington
Locations (1):
- Missouri Breaks Industries Research Inc, Eagle Butte, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hawley CN, Huber CM, Best LG, Howard BV, Umans J, Beresford SAA, McKnight B, Hager A, O'Leary M, Thorndike AN, Ornelas IJ, Brown MC, Fretts AM. Cooking for Health: a healthy food budgeting, purchasing, and cooking skills randomized controlled trial to improve diet among American Indians with type 2 diabetes. BMC Public Health. 2021 Feb 15;21(1):356. doi: 10.1186/s12889-021-10308-8. PMID 33588808

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant events after participant enrollment, but prior to randomization to intervention or control arm.
Groups:
- Control Arm: No intervention (all intervention materials were given to participants randomized to the control arm at the end of the study)
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 88 | 88
Month 6 Visit | 74 | 79
Completed | 71 | 82
Not Completed | 17 | 6
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 10 | 3
Not completed — Withdrawal by Subject | 5 | 0
Not completed — incarcerated | 1 | 0
Not completed — scheduled, but no show | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 88 | 88 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (11.9) | 48.3 (11.2) | 49.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 58 | 127
  Male | 19 | 30 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 88 | 88 | 176
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Sugar-sweetened beverages [Mean (Standard Deviation); unit: servings per day] | 1.2 (2.4) | 1.1 (1.6) | 1.2 (2.0)
Unhealthy Food Purchases [Mean (Standard Deviation); unit: purchases per 30 days] | 39.4 (34.7) | 51.2 (38.2) | 45.3 (36.8)
Healthy Food Purchases [Mean (Standard Deviation); unit: purchases per 30 days] | 62.4 (56.0) | 88.0 (75.2) | 75.3 (67.4)

OUTCOME MEASURES:

1. Primary Outcome: Change (From Baseline) in Self-reported Intake (Servings/Day) of Sugar-sweetened Beverages (Measured Using the Nutrition Assessment Shared Resource Food Frequency Questionnaire) at 6 Months and 12 Months
Description: Sugar-sweetened beverages include self-reported intake of fruit drinks, sugar-based energy drinks, and soda. Intake of sugar-sweetened beverages will be estimated using measures of consumption frequency and portion size. Average intakes will be calculated for each study participant using the University of Minnesota Nutrition Data Systems for Research Software by multiplying the frequency response for each beverage on the food frequency questionnaire by the recalled portion size, and then summing for all relevant beverages. Change from baseline with be assessed at 6 months and 12 months (12 months - baseline; 6 months - baseline). As the intervention hopes to decrease intake of sugar-sweetened beverages, lower (i.e., more negative) after - before differences represent a better outcome.
Time Frame: measured at baseline, and months 6 and 12
Population: Participants who completed the food frequency questionnaire at the baseline and month 6 exam or the baseline and month 12 exam
Measure: Mean (Standard Error); unit: servings
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 70 | 78
servings
  12 months-baseline: number analyzed (Participants) | 67 | 78
  12 months-baseline | -0.13 (0.38) | -0.11 (0.28)
  6 months-baseline: number analyzed (Participants) | 70 | 75
  6 months-baseline | -0.22 (0.23) | -0.28 (0.21)

2. Primary Outcome: Change (From Baseline) in Healthy and Unhealthy Food Purchases (Measured Using the Healthy/Unhealthy Food Acquisition Survey) at 6 Months and 12 Months
Description: Change in healthy and unhealthy food purchases will be estimated using the Healthy/Unhealthy Food Acquisition Survey. The survey includes a list of 47 healthy and unhealthy foods commonly consumed in the community. At each exam (baseline, month 6, month 12), participants will report the number of times he/she acquired each of the 47 foods in the past 30 days. Change from baseline with be assessed at 6 months and 12 months (12 months - baseline; 6 months - baseline). As the intervention hopes to increase the number of healthy food purchases and decrease the number of unhealthy food purchases, higher after - before differences represent a better outcome for healthy foods and lower after - before differences represent a better outcome for unhealthy foods.
Time Frame: measured at baseline, and months 6 and 12
Population: Participants who completed the healthy and unhealthy food purchases questionnaire at the baseline and month 6 exam or the baseline and month 12 exam
Measure: Mean (Standard Error); unit: purchases per 30 days
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 72 | 82
purchases per 30 days
  12 months-baseline, unhealthy food purchases: number analyzed (Participants) | 69 | 82
  12 months-baseline, unhealthy food purchases | -7.4 (3.3) | -10.1 (3.7)
  6 months-baseline, unhealthy food purchases: number analyzed (Participants) | 72 | 79
  6 months-baseline, unhealthy food purchases | -6.42 (4.92) | -9.91 (4.25)
  12 months-baseline, healthy food purchases: number analyzed (Participants) | 70 | 82
  12 months-baseline, healthy food purchases | 7.24 (4.95) | -16.3 (8.56)
  6 months-baseline, healthy food purchases: number analyzed (Participants) | 72 | 78
  6 months-baseline, healthy food purchases | 0.84 (6.3) | -10.5 (0.84)

3. Secondary Outcome: Change (From Baseline) in Food Budgeting Skills (Measured Using the Food Resource Management Scale) at 6 Months and 12 Months
Description: Change in food budgeting skills will be estimated using the Food Resource Management Scale. The scale includes 4 questions related to shopping behaviors to maximize food resources. The Food Resource Management Scale is a Likert-type scale with responses ranging from 1 (never) to 5 (always). Responses to the four questions will be averaged to create a total Food Resource Management Score. Change from baseline with be assessed at 6 months and 12 months (12 months - baseline; 6 months - baseline). As the intervention hopes to increase food budgeting skills, higher after-before differences represent a better outcome.
Time Frame: measured at baseline, and months 6 and 12
Population: Participants who completed the Food Resource Management questions at the baseline and month 6 exam or the baseline and month 12 exam
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 73 | 80
score on a scale
  12 months-baseline: number analyzed (Participants) | 69 | 80
  12 months-baseline | 0.28 (0.11) | -0.08 (0.10)
  6 months-baseline: number analyzed (Participants) | 73 | 77
  6 months-baseline | 0.08 (0.12) | 0.05 (0.10)

4. Secondary Outcome: Change (From Baseline) in Cooking Skills (Measured Using the Cooking Confidence Scale) at 6 Months and 12 Months
Description: Change in cooking skills will be estimated using a minor modification of the Cooking Confidence Scale. The Cooking Confidence Scale includes 6 questions related to confidence in preparing healthy foods. It is a Likert-type scale with responses ranging from 1 (not at all confident) to 5 (very confident). Responses to the questions will be averaged. Change from baseline with be assessed at 6 months and 12 months (12 months - baseline; 6 months - baseline). As the intervention hopes to increase cooking skills, higher after - before differences represent a better outcome.
Time Frame: measured at baseline, and months 6 and 12
Population: Participants who completed the Cooking Confidence Scale questions at the baseline and month 6 exam or the baseline and month 12 exam
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 68 | 78
score on a scale
  12 months-baseline: number analyzed (Participants) | 64 | 78
  12 months-baseline | 0.16 (0.08) | -0.18 (0.09)
  6 months-baseline | 0.21 (0.06) | -0.06 (0.08)

5. Secondary Outcome: Process Evaluation: Intervention Reach
Description: The proportion of those approached that were eligible for the intervention (and the number who subsequently participate) will be used as a marker of intervention reach.
Time Frame: Years 2020-2023
Reporting Status: Not Posted

6. Secondary Outcome: Process Evaluation: Intervention Fidelity
Description: The investigators will assess adherence to the study protocol and document barriers and facilitators to implementation throughout the trial.
Time Frame: through study completion, estimated 12 months to complete intervention per participant
Reporting Status: Not Posted

7. Secondary Outcome: Process Evaluation: Intervention Satisfaction (Among Those in the Intervention Arm)
Description: During months 6 and 12, a sub-sample of study participants in the intervention arm will meet with study staff by phone for semi-structured interviews to evaluate the overall intervention. Qualitative analyses will assess participant's satisfaction with the intervention.
Time Frame: Semi-structured interviews will be done at months 6 and 12.
Reporting Status: Not Posted

8. Secondary Outcome: Process Evaluation: Intervention Dose Delivered (i.e., Number of Lessons Included in the Curriculum Available for Participants)
Description: Dose will be assessed in the intervention arm only
Time Frame: through study completion, estimated 12 months to complete intervention per participant
Reporting Status: Not Posted

9. Secondary Outcome: Process Evaluation: Intervention Dose Received (i.e., Number of Lessons Included in the Curriculum Completed by Participants)
Description: Dose will be assessed in the intervention arm only
Time Frame: through study completion, estimated 12 months to complete intervention per participant
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the one year (baseline through month 12 visit).
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 1/88 | 2/88
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/88
Other Adverse Events (participants affected / at risk) | 0/88 | 0/88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT03699709/Prot_SAP_000.pdf